CLINICAL TRIAL: NCT05994742
Title: Co-SAM: An Adaptive Multi-arm Trial to Improve Clinical Outcomes Among Children Recovering From Complicated Severe Acute Malnutrition
Brief Title: An Adaptive Multi-arm Trial to Improve Clinical Outcomes Among Children Recovering From Complicated SAM
Acronym: Co-SAM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Oxford (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); University of Washington (Other); Wageningen University (Other); Zvitambo Institute for Maternal & Child Health (Unknown); Tropical Gastroenterology & Nutrition Group (TROPGAN) (Other); University of Cambridge (Other); Kenya Medical Research Institute (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150522
Record Dates: First submitted 2023-07-14; First posted 2023-08-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Severe Acute Malnutrition; HIV; Comorbidities and Coexisting Conditions; Child Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition; Child Nutrition Disorders | interventions — Rifampin; Azithromycin; Isoniazid; Pyridoxine; Child Development; Standard of Care

STUDY DESIGN:
Intervention Model Description: Adaptive, multi-arm randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1: Standard-of-care (control) (Active Comparator): Children in the control arm will receive Ready to Use Therapeutic Food (RUTF) for at least 2 weeks, plus all standard care. Children with HIV will receive long-term Cotrimoxazole prophylaxis and antiretroviral therapy, as per current guidelines.
  Interventions: Other: Standard Care
- Arm 2: Antimicrobial package (Experimental): Children will receive a bundle of azithromycin (3 days every month), isoniazid (daily), rifampicin (daily) and pyridoxine (daily) for 12 weeks.
  Interventions: Drug: Rifampicin; Drug: Azithromycin; Drug: Isoniazid; Drug: Pyridoxine Hydrochloride; Other: Standard Care
- Arm 3: Reformulated RUTF (Experimental): Children will receive a reformulated RUTF, with increased medium-chain triglycerides (MCTs), higher hydrolysed protein content and a more bioavailable form of selenium (selenium yeast). Children will receive RUTF for at least 2 weeks.
  Interventions: Dietary Supplement: Reformulated Ready to Use Therapeutic Food; Other: Standard Care
- Arm 4: Psychosocial package (Experimental): Caregiver-child pairs will receive a low-cost, co-designed intervention to strengthen caregiver support, enhance income generation and promote child play. This is delivered over 12 weeks and comprises:
  i) The Friendship Bench, developed as a low-cost psychological intervention utilising problem-solving therapy (delivered by trained lay workers) and peer-to-peer support to address depression and other common mental disorders.
  ii) Care for Child Development is a UNICEF package that helps families build stronger relationships and solve problems in caring for the child at home, through play and communication activities in a series of age-appropriate interactive modules delivered by a lay worker using 'flash' cards.
  iii) Educational and behaviour-change messages around better nutrition; play for children with SAM; stigma, HIV and gender-based violence; financial planning; causes of SAM; and health-seeking behaviours.
  Interventions: Behavioral: The Friendship Bench; Behavioral: Care for Child Development; Behavioral: Educational and behaviour-change modules; Other: Standard Care
- Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package (Experimental): A combination of all interventions from arms 2, 3 and 4, plus standard care delivered for 12 weeks.
  Interventions: Drug: Rifampicin; Drug: Azithromycin; Drug: Isoniazid; Drug: Pyridoxine Hydrochloride; Behavioral: The Friendship Bench; Behavioral: Care for Child Development; Behavioral: Educational and behaviour-change modules; Dietary Supplement: Reformulated Ready to Use Therapeutic Food; Other: Standard Care

INTERVENTIONS:
Drug: Rifampicin — Rifampicin is commonly used in the first-line management of paediatric tuberculosis, and is approved by the FDA (ID: 2862628) and the EMA (EMA/31710/2020).
  Arms: Arm 2: Antimicrobial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Drug: Azithromycin — Azithromycin is a macrolide antibiotic, and is approved for use in children by the FDA (ID: 3263750) and EMA (EMA/2872/2021).
  Arms: Arm 2: Antimicrobial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Drug: Isoniazid — Isoniazid is an antibiotic commonly used in the firstline treatment of tuberculosis, and as tuberculosis prophylaxis.
  Arms: Arm 2: Antimicrobial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Drug: Pyridoxine Hydrochloride — Pyridoxine is a form of vitamin B6 used to prevent peripheral neuropathy among children receiving isoniazid.
  Arms: Arm 2: Antimicrobial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Behavioral: The Friendship Bench — The Friendship Bench was developed in Zimbabwe as a low-cost psychological intervention utilising problemsolving therapy (delivered by trained lay workers) and peer-to-peer support to address depression and other common mental disorders. There is a strong evidence base for its use in urban LMIC settings. Peer support groups meet every 1-2 weeks and focus on communal problem solving, and establishing income-generation activities (such as making bags).
  Arms: Arm 4: Psychosocial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Behavioral: Care for Child Development — Care for Child Development is a UNICEF package that helps families build stronger relationships and solve problems in caring for the child at home, through play and communication activities to stimulate children, through a series of age-appropriate interactive modules delivered by a lay worker using 'flash' cards. It has been used in other African contexts and has good acceptability.
  Arms: Arm 4: Psychosocial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Behavioral: Educational and behaviour-change modules — Educational and behaviour-change messages around better nutrition; play for children with SAM; stigma,HIV and gender-based violence; financial planning; causes of SAM; and health-seeking behaviours. These have been developed with caregivers affected by SAM in a previous study, through a series of codesign workshops, ensuring these are contextually relevant.
  Arms: Arm 4: Psychosocial package; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Dietary Supplement: Reformulated Ready to Use Therapeutic Food — A reformulated product designed to improve outcomes for children who have severe acute malnutrition.
  Arms: Arm 3: Reformulated RUTF; Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package
Other: Standard Care — All children will receive care according to WHO guidelines, which includes standard RUTF and any other medications required.

SUMMARY:
Malnutrition underlies 45% of child deaths, and has far-reaching educational, economic and health consequences. Severe acute malnutrition (SAM) affects 17 million children globally and is the most life-threatening form of malnutrition. Community-based management of acute malnutrition using ready-to-use therapeutic food (RUTF) has transformed outcomes for children with uncomplicated SAM, but those presenting with poor appetite or medical complications (categorised as having 'complicated' SAM) require hospitalisation. Data show that pneumonia, diarrhoea and malaria are leading causes of death in children with complicated SAM after discharge from hospital. High risk of infectious deaths suggests that sustained antimicrobial interventions may reduce mortality following discharge from hospital. Furthermore, children with complicated SAM respond less well to nutritional rehabilitation, and oftentimes are discharged to a home environment characterised by poverty and multiple caregiver vulnerabilities including depression, low decision making autonomy, lack of social support, gender-restricted family relations, and competing demands on scarce resources. Caregivers have to navigate diverse challenges that impede engagement with clinical care after discharge from hospital. The objective is to address the biological and social determinants of multimorbidity in children with complicated SAM by developing multimodal packages of interventions and testing them in a 5-arm adaptive randomized controlled clinical trial, with death/hospitalization or failed nutritional recovery as the primary outcome.

DETAILED DESCRIPTION:
This is a 5-arm randomized, unblinded clinical trial comparing:

Arm 1: Standard-of-care (control) Arm 2: Antimicrobial package Arm 3: Reformulated RUTF Arm 4: Psychosocial package Arm 5: Antimicrobial package + reformulated RUTF + psychosocial package

The trial will test the superiority of each intervention arm over the standard of care arm (control). Children in the control arm (and all intervention arms) will receive RUTF for at least 2 weeks and all standard care. The trial is adaptive, meaning i) that each intervention arm will be added as it becomes available, and ii) an interim analysis will enable us to drop arms which are unpromising based on pre-specified criteria. There will be no blinding or placebo, because the very different components in each trial arm make it very challenging to blind. Children with complicated SAM will be screened and enrolled from hospital sites shortly before discharge, and interventions will be started before leaving hospital, and continued for 12 weeks through outpatient visits. Children will be followed at 2, 4, 6, 8, 12 and 24 weeks post-discharge in dedicated study clinics (with additional visits at 1, 3 and 5 weeks for caregiver-child pairs receiving the psychosocial intervention).

The primary outcome is death or hospitalization or failed nutritional recovery by 24 weeks.

The aim is to recruit 1266 children across three countries. The study is not testing new drugs but rather testing a different package of medications (Arms 2 and 5) as compared to current standard care, which the investigator believe will have greater benefit. The RUTF will be a new formula in two of the arms (3 and 5) based on research into what composition will improve health outcomes for children with complicated SAM. This will be a variant on Plumpy'Nut®, a brand that is known and trusted, produced in collaboration with the manufacturers, Nutriset.

The Psychosocial intervention (Arms 4 and 5) will involve three components:

i) The Friendship Bench, which was developed in Zimbabwe as a low-cost psychological intervention utilising problem-solving therapy (delivered by trained lay workers) and peer-to-peer support to address depression and other common mental disorders. There is a strong evidence-base for its use in urban LMIC settings. Peer support groups meet every 1-2 weeks and focus on communal problem solving, and establishing income-generation activities (such as making bags). ii) Care for Child Development is a UNICEF package that helps families build stronger relationships and solve problems in caring for the child at home, through play and communication activities to stimulate children, through a series of age-appropriate interactive modules delivered by a lay worker using 'flash' cards. It has been used in other African contexts and has good acceptability. iii) Educational and behavior-change messages around better nutrition; play for children with SAM; stigma, HIV and gender-based violence; financial planning; causes of SAM; and health-seeking behaviours.

Blood and stool will be collected at baseline, 12 and 24 weeks from all children to explore recovery of underlying pathological processes. At week 2, liver function tests will be undertaken in local laboratories. Samples will also be transported to Kenya and the Netherlands for some assays not available in each country.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months, of either sex
* Hospitalised with complicated severe acute malnutrition, as per WHO definition
* Started transition to RUTF
* Caregiver willing and able to attend the study clinic for all visits
* Caregiver able and willing to give informed consent

Exclusion Criteria:

* Any acute or chronic condition which mean that receipt of one or more study interventions, or participation in the trial, would not be advisable.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1266 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Death or first hospitalisation or failed nutritional recovery within 24 weeks post-randomisation | 24 weeks post-randomisation
  a) All-cause mortality. b) Overnight admission to a health facility for any reason. This includes cases where there was a clinical plan to hospitalise the child, which was refused by the caregiver. c) Failed nutritional recovery is defined as either: i) Persistent WHZ<-2 or MUAC<12.5cm or bilateral pedal oedema at week 12; or ii) WHZ<-2 or MUAC<12.5cm or bilateral pedal oedema at any time between baseline and week 24 post-randomisation in a child who had previously recovered.

SECONDARY OUTCOMES:
Change in weight-for-height Z-score | 24 weeks post-randomisation
  Change in weight-for-height Z-score between baseline and 24 weeks post-randomisation according to age- and-sex appropriate WHO reference standards.
Change in mid-upper arm circumference | 24 weeks post-randomisation
  Change in size of mid-upper arm in centimetres between baseline and 24 weeks.
Change in weight-for-age Z-score | 24 weeks post-randomisation
  Change in weight-for-age Z-score between baseline and 24 weeks post-randomisation according to age- and sex-appropriate WHO reference standards.
Change in height-for-age Z-score | 24 weeks post-randomisation
  Change in height-for-age Z-score between baseline and 24 weeks post-randomisation according to age- and sex-appropriate WHO reference standards.
Number of participants with suspected or confirmed tuberculosis,pneumonia, diarrhoea or malaria | 24 weeks post-randomisation
  Physician-diagnosed suspected or confirmed infection, as defined by WHO guidelines, between baseline and 24 weeks post-randomisation.

OTHER OUTCOMES:
Change in anthropometry: Weight-for-height Z score (WHZ) | 4 weeks post-randomisation and 12 weeks post-randomisation
  Change in WHZ between baseline and 4 weeks post-randomisation, and baseline and 12 weeks post-randomisation.
Change in anthropometry: Weight-for-age Z score (WAZ) | 4 weeks post-randomisation and 12 weeks post-randomisation
  Change in WAZ between baseline and 4 weeks post-randomisation, and baseline and 12 weeks post-randomisation.
Change in anthropometry: Height-for-age Z score (HAZ) | 4 weeks post-randomisation and 12 weeks post-randomisation
  Change in HAZ between baseline and 4 weeks post-randomisation, and baseline and 12 weeks post-randomisation.
Change in anthropometry: Mid-upper arm circumference (MUAC) | 4 weeks post-randomisation and 12 weeks post-randomisation
  Change in MUAC between baseline and 12 weeks post-randomisation.
Change in caregiver mental health | 24 weeks post-randomisation
  Change in Shona Symptom Questionnaire score (and proportion meeting cut-off score >8) between baseline and 24 weeks post-randomisation. This is a widely used 10-item self-report questionnaire. Each item is scored from 0-3, leading to a total score between 0-30, with higher scores indicating more severe depressive symptoms.
Concentration of lipid mediators/proteins | 12 weeks and 24 weeks post-randomisation
  LC-MS measurement of fatty acids, acylcarnitines, polyamines, amino acids, glycolysis intermediates, TCA cycle intermediates, nucleotides, prostaglandins, serotonin, bile acids, lysophosphatidylcholines, phosphatidylcholines, cholesterol and derivatives, organic acids and tri/di/monoglycerides.
Concentration of metabolites | 12 weeks and 24 weeks post-randomisation
  Luminex measurement of Insulin, Insulin-like growth factor 1, leptin, ghrelin, cortisol, growth hormone, Glucagon-like peptide-1, Peptide YY, Monocyte chemoattractant protein-1, and Plasminogen activator inhibitor-1.
Concentration of inflammatory mediators | 12 weeks and 24 weeks post-randomisation
  Luminex measurement of chemokines, cytokines and circulating growth factors.

CONTACTS AND LOCATIONS:
Locations (5):
- Zambia (2):
  - Matero Hospital, Lusaka
  - UTH - University Teaching Hospital, Lusaka
- Zimbabwe (3):
  - Chitungwiza Central Hospital, Harare
  - Parirenyatwa Hospital, Harare
  - Sally Mugabe Hospital, Harare

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at the end of the trial on ClinEpiDB.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2028
Access Criteria: Via ClinEpiDB
URL: http://clinepidb.org

REFERENCES:
- [Derived] Bwakura-Dangarembizi M, Amadi B, Singa BO, Muyemayema S, Ngosa D, Mwalekwa L, Ngao N, Kazhila L, Mutasa B, Mpofu E, Mudawarima L, Gonzales GB, Mudzingwa S, Mutenda M, Keter LK, Mutasa K, Njunge JM, Jones H, Phiri TN, Mudibo E, Chulu N, Majo FD, Chasekwa B, Tembo A, Nyabinda C, Oduol C, Sauramba V, Tavengwa NV, Langhaug L, Cordani I, Smuk M, Jaki T, Ntozini R, Walson J, Tickell KD, Berkley J, Kelly P, Prendergast AJ; Co-SAM Trial Team. An adaptive multiarm randomised trial of biomedical and psychosocial interventions to improve convalescence following severe acute malnutrition in sub-Saharan Africa: Co-SAM trial protocol. BMJ Open. 2025 May 24;15(5):e093758. doi: 10.1136/bmjopen-2024-093758. PMID 40413053